CLINICAL TRIAL: NCT05930314
Title: CNCT19 Cell Injection for Refractory Systemic Lupus Erythematosus
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001009
Record Dates: First submitted 2023-06-24; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Refractory Systemic Lupus Erythematosus; Lupus Nephritis; Immune Thrombocytopenia
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: refractory systemic lupus erythematosus(SLE) presented with active lupus nephritis or active immune thrombocytopenia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNCT19 cell injetion (Experimental): CNCT19 administration：0.25 to 0.5 x 10^8 CAR-positive viable
  Interventions: Drug: CNCT19 cell injection

INTERVENTIONS:
Drug: CNCT19 cell injection — Leukapheresis and manufacturing of CNCT19: enrolled subjects will undergo a leukapheresis to target a yield of > 1x 10^9 mononuclear cells
  * Lymphodepleting chemotherapy i. Fludarabine 25 to 30 mg/m2, once daily for 3 days ii. Cyclophosphamide 500 mg/m2, once daily for 3 days
  * CNCT19 administration i. 0.25 to 0.5 x 10^8 CAR-positive viable T cells

SUMMARY:
Investigator-initiated, single-arm, open-label, single dose clinical study to evaluate the safety and preliminary efficacy of CNCT19 in treatment of patients with refractory systemic lupus erythematosus(SLE) presented with active lupus nephritis or active immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to sign Informed Consent Form (ICF) ;
* 2. Males or females 18-70（include 18 and 70） years of age;
* 3. Have a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) 1997 or European League against Rheumatism(EULAR)/ the American College of Rheumatology (ACR) 2019 criteria .Have a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) 1997 or European League against Rheumatism(EULAR)/ the American College of Rheumatology (ACR) 2019 criteria .

Group1:Have active, biopsy-proven proliferative lupus nephritis Class III or IV, or Class V using the 2003 ISN/RPS criteria. The biopsy must be performed in the 6 months prior to the screening visit or during the screening period. Have documentation of active renal disease defined as:24h Proteinuria> 1.5 grams/day.

Refractory lupus nephritis is defined as no induced remission to treatment regimens containing at least one immunosuppressant (including glucocorticoids, CTX, tacrolimus, MMF, and cyclosporine) after 3 to 6 months, accompanied by no reduction (or worsening) of proteinuria or persistent antibody positives.

Group 2: Refractory thrombocytopenia: No response to treatment with at least 1 course of MP shock (1g for 3 days) or high dose of glucocorticoids (1mg/kgd equivalent dose of glucocorticoids) combined with 1 or more immunosuppressants. Before enrollment, at least 2 consecutive blood routine tests were performed to check platelets below 50×10^9/L and above 30×10^9/L. Other non-SLE causes of thrombocytopenia, such as infection, bone marrow suppression, and hypersplenism, were excluded.

* 4. Not pregnant or nursing.
* 5. Adequate organ functions indicated as: ALT and AST < 3 times of the ULN； Total bilirubin < 2mg/dL with the exception of patients with Gibert-Meulengracht syndrome, who may be included if their total bilirubin is < 3 x ULN and direct bilirubin < 1.5mg/dL ULN； An estimated glomerular filtration rate < 30 mL/min/1.73 m^2 at the screening visit Serum creatinine ≤1.5mg/dl(133umol/l); Must have a minimum level of pulmonary reserve, non-oxygenated blood oxygen saturation >95%;
* 6. Lymphocyte count > 0.4×10^9/L；
* 7. Use a small dose of glucocorticoid (dose equivalent to ≤10mg/d prednisone) for not less than 1 month (except glucocorticoid intolerance).

Exclusion Criteria:

* 1. Severe active central nervous system (CNS) lupus, including seizures, psychosis, cerebrovascular accidents;
* 2. Dialysis patients or creatinine clearance rate < 30ml/min；
* 3. Pregnant or breast feeding；
* 4. Active infections (such as sepsis, bacteremia, fungemia, uncontrolled pulmonary infection, and active tuberculosis);
* 5. One of the following: HBsAg positive HCV-Ab positive HIV positive TP positive
* 6. Undergone major surgery assessed by the subjects as unsuitable for inclusion within 4 weeks prior to screening.
* 7. Had or is currently suffering from other malignant tumors within five years prior to screening, except for curable tumors with negligible risk of metastasis or death, such as cervical carcinoma in situ and skin basal cell carcinoma with adequate treatment;
* 8. The heart meets any of the following conditions: Left ventricular ejection fraction (LVEF) ≤45%; New York Heart Association (NYHA) Class III or IV congestive heart failure or active heart disease; Severe arrhythmias requiring treatment (except atrial fibrillation and paroxysmal supraventricular tachycardia); QTcB interval male ≥450ms, female ≥470ms (QTcB=QT/RR^1/2); Had a myocardial infarction, bypass, or stent surgery within the 6 months prior to the study; Other heart diseases that the investigators judged unsuitable for inclusion;
* 9. Received live vaccine within 6 weeks prior to screening；
* 10. Participants who have participated in other interventional clinical studies within the 3 months prior to cell transfusion, received active investigational drug therapy, or who intend to participate in another clinical trial or receive treatment outside the protocol during the entire study period.
* 11. a history of epilepsy or other active central nervous system diseases;
* 12. Subjects who are known to have hypersensitivity to the ingredients of the preparation used in the test;
* 13. Previously received CAR T cell therapy;
* 14. Other conditions deemed unsuitable for participation in this clinical trial by subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Dr, Principal Investigator — Peking Union Medical College Hospital; Daobin Zhou, Dr, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Xiaofeng Zeng, Beijing, China